CLINICAL TRIAL: NCT00811473
Title: An 8-week, Multicenter, Double-blind, Randomized, Parallel-group, Placebo-controlled Study of the Efficacy and Safety of Quetiapine Fumarate (SEROQUEL) Extended-Release in Children and Adolescent Subjects With Bipolar Depression
Brief Title: Pediatric Bipolar Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D144AC00001
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2011-12-01 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Bipolar Depression
Keywords: Bipolar Depression; Depression; Children; Adolescents; Seroquel; Bipolar Depression in Children and Adolescents
MeSH Terms: conditions — Bipolar Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Quetiapine XR (Experimental)
  Interventions: Drug: Quetiapine XR
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine XR — Oral treatment with 150 up to 300 mg/day once daily in the evening
  Other Names: Seroquel XR
  Arms: Quetiapine XR
Drug: Placebo — Oral treatment once daily in the evening
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if quetiapine fumarate extended-release (quetiapine XR or SEROQUEL® XR) 150 to 300 mg/day taken by itself is effective and safe in treating children or adolescents aged 10 to 17 with bipolar depression and if so, how it compares with placebo (a non-active tablet, like a sugar pill, that looks like quetiapine).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent by one or both parents or legal guardian and written assent by the patients before any study procedures are performed.
* The patient must have a documented clinical diagnosis for bipolar I or bipolar II disorder, and including current episode depressed.
* Patients are required to be in outpatient status at the enrollment and randomization visits and believed likely to remain an outpatient for the duration of the study.
* Patients must be able to swallow the study medication tablets.

Exclusion Criteria:

* The patient must not have been diagnosed with Tourette's Disorder, Obsessive-Compulsive Disorder, acute Post-traumatic Stress Disorder, Panic Disorder, Autistic Disorder and/or Asperger's Disorder.
* Patient can not have a history of non-response to an adequate treatment to more than 2 antidepressants during the current episode.
* The patient must not have received electroconvulsive therapy (ECT) within 30 days before participating in the study.
* Patients who in your doctors judgement pose a current suicidal or homicidal risk.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 193 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Castiglione, Study Director — AstraZeneca; Robert L. Findling, Principal Investigator — University Hospitals Case Medical CenterCase Western Reserve University School of Medicine
Locations (48):
- United States (31):
  - Research Site, Dothan, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Escondido, California
  - Research Site, Bradenton, Florida
  - Research Site, Gainsville, Florida
  - Research Site, North Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Smyrna, Georgia
  - Research Site, Eagle, Idaho
  - Research Site, Hoffman Estates, Illinois
  - Research Site, Terre Haute, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Clinton Township, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Flowood, Mississippi
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Rochester, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Mason, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Wharton, Texas
  - Research Site, Virginia Beach, Virginia
  - Research Site, Bothell, Washington
  - Research Site, Milwaukee, Wisconsin
- Colombia (4):
  - Research Site, Bogota D.c, Cundinamarca
  - Research Site, Bello
  - Research Site, Bogotá
  - Research Site, Medellín
- India (4):
  - Research Site, Vijaywada, Andh Prad
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Varanasi, Uttar Prad
- Mexico (2):
  - Research Site, León
  - Research Site, Monterrey
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Novi Sad
- South Africa (2):
  - Research Site, Pretoria, Gauteng
  - Research Site, Cape Town, W Cape
- Taiwan (3):
  - Research Site, Taoyuan District, Taiwan
  - Research Site, Changhua
  - Research Site, Taipei

REFERENCES:
- [Background] Findling RL, Pathak S, Earley WR, Liu S, DelBello MP. Efficacy and safety of extended-release quetiapine fumarate in youth with bipolar depression: an 8 week, double-blind, placebo-controlled trial. J Child Adolesc Psychopharmacol. 2014 Aug;24(6):325-35. doi: 10.1089/cap.2013.0105. Epub 2014 Jun 23. PMID 24956042
- See also: CSR-D144AC00001.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=276&filename=CSR-D144AC00001.pdf
- See also: D144AC00001_Redacted_Study_Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=276&filename=D144AC00001_Redacted_RRB_1516423827582625983.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted between 27 January 2009 and 1 November 2010, which included the recall visit. The recall visit occurred from 5 June 2010 till 1 November 2010.
Pre-assignment Details: The study had an up to 35-day enrollment period, 8-week double-blind treatment period with 1 of 2 treatment regimens (quetiapine XR 150 to 300 mg/day or placebo), 1-week safety follow-up period, 2- to 4-week safety follow-up period for patients with BP >95th percentile at completion/discontinuation.
Groups:
- Quetiapine XR: Quetiapine XR 150 to 300mg once a day
- Placebo: Matching placebo
Period: Overall Study
Arm/Group | Quetiapine XR | Placebo
Started | 93 | 100
Completed | 70 | 74
Not Completed | 23 | 26
Not completed — Adverse Event | 3 | 12
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Severe non-compliance to protocol | 2 | 4
Not completed — Lack of therapeutic response | 4 | 1
Not completed — Condition under investigation worsened | 1 | 3
Not completed — Other 2 | 4 | 1
Not completed — Incorrect Enrollment | 1 | 0
Not completed — Safety Reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine XR | Placebo | Total
Number analyzed (Participants) | 92 | 100 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety analysis set
  years | 13.9 (2.18) | 14.0 (2.05) | 14.0 (2.11)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety analysis set
  Participants
    Female | 47 | 48 | 95
    Male | 45 | 52 | 97

OUTCOME MEASURES:

1. Primary Outcome: Change in the Children Depression Rating Scale, Revised (CDRS-R) Total Score From Baseline to Final Assessment (Day 57)
Description: Severity of depression in children and adolescents was calculated based on the 17-item CDRS-R scale (3 items scored from 1-5 and 14 items scored from 1-7, with higher scores indicating more severe depression). The 17 item scores are summed to give the total score (total score range 17-113).
Time Frame: Will be scored at all visits. the analysis is the change from baseline to the final assessment at day 57
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 92 | 100
Scores on a scale | -29.6 (1.65) | -27.3 (1.60)

2. Secondary Outcome: Number of Patients Reaching Remission Where Remission is Defined as CDRS-R Total Score ≤28 at Final Assessment (Day 57).
Description: The number of patients with remission from Days 8 to 57 was calculated. The CDRS-R is a 17-item scale with 3 items scored from 1-5 and 14 items scored from 1-7, where higher scores indicating more severe depression. The 17 item scores are summed to give the total score (total score range 17-113).
Time Frame: Days 8 to 57
Measure: Number; unit: participants
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 92 | 100
participants | 42 | 34

3. Secondary Outcome: The Number of Patients With the Response, Where Response is Defined as ≥50% Reduction From Baseline to Final Assessment (Day 57) in CDRS-R Total Score
Description: The number of patients reaching response from Days 8 to 57 was calculated. The CDRS-R is a 17-item scale with 3 items scored from 1-5 and 14 items scored from 1-7, where higher scores indicating more severe depression. The 17 item scores are summed to give the total score (total score range 17-113).
Time Frame: Days 8 to 57
Measure: Number; unit: participants
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 92 | 100
participants | 58 | 55

4. Secondary Outcome: Change From Baseline to Final Assessment (Day 57) in the CGI-BP-S
Description: The CGI-BP-S scale rates the severity of the patient's illness at the time of assessment and is scored from 1 to 7 (1=normal, not ill to 7=very severely ill). Higher CGI-BP-S scores indicate greater illness severity.
Time Frame: Change from Baseline to Day 57
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 92 | 100
Scores on a Scale | -17.2 (0.15) | -1.35 (0.14)

5. Secondary Outcome: CGI-BP-C Score at Final Assessment (Day 57)
Description: The CGI-BP-C scale rates how much the patient's illness has improved or worsened compared to the phase immediately preceding treatment and is scored on a scale from 1 to 8 (1=very much improved to 7=very much worse; 8=not applicable). CGI-BP-C scores >4 indicate worsening, while scores <4 indicate improvement.
Time Frame: Change from Baseline to day 57
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 92 | 100
Scores on a scale | 2.4 (0.15) | 2.6 (0.15)

6. Secondary Outcome: The Proportion of Patients at Final Assessment (Day 57) With Improvement of Overall Bipolar Illness
Description: The proportion of patients with improvement of overall bipolar illness at Day 57 was calculated. Improvement defined as a CGI-BP-C of "Much" or "Very much" improved in overall bipolar illness assessment.
Time Frame: Day 57
Measure: Number; unit: Proportions
Arm/Group | Quetiapine XR | Placebo
Number analyzed (Participants) | 92 | 100
Proportions | 0.522 | 0.40

ADVERSE EVENTS:
Arm/Group | Quetiapine XR | Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 4
Other Adverse Events (participants affected / at risk) | 68/92 | 66/100
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Quetiapine XR | Placebo
Agitation (Psychiatric disorders) | 1/92 | 0/100
Social Stay Hospitalisation (Social circumstances) | 0/92 | 1/100
Bipolar Disorder (Psychiatric disorders) | 0/92 | 1/100
Aggression (Psychiatric disorders) | 0/92 | 1/100
Depressive Symptoms (Psychiatric disorders) | 0/92 | 1/100
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR (N=92) | Placebo (N=100)
Headache (Nervous system disorders) | 20 | 12
Sedation (Nervous system disorders) | 7 | 6
Dizziness (Nervous system disorders) | 6 | 2
Somnolence (Nervous system disorders) | 6 | 4
Influenza (Infections and infestations) | 4 | 1
Nasoparyngitis (Infections and infestations) | 4 | 3
Gastroenteritis (Infections and infestations) | 3 | 0
Sinusitis (Infections and infestations) | 3 | 0
Urinary Tract Infection (Infections and infestations) | 3 | 0
Ear Infection (Infections and infestations) | 2 | 0
Upper respiratory Tract Infection (Infections and infestations) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Nausea (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3
Abdominal Pain (Gastrointestinal disorders) | 2 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 5 | 2
Irritability (General disorders) | 2 | 5
Pyrexia (General disorders) | 2 | 1
Thirst (General disorders) | 2 | 0
Influenza like illness (General disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 0
Nightmare (Psychiatric disorders) | 2 | 2
Aggression (Psychiatric disorders) | 0 | 2
Increased Appetite (Metabolism and nutrition disorders) | 3 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 2
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 | 1
Orthodontic Appliance Complication (Injury, poisoning and procedural complications) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days